CLINICAL TRIAL: NCT01903824
Title: A Double-Blind, Placebo- and Positive-Controlled, Randomized, Partial 6-way Crossover Study to Investigate the Pharmacodynamics and Pharmacokinetics of CEP-26401 (5, 25, and 125 μg) Following Single-Dose Administration to Healthy Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics (PK/PD) of CEP-26401 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: C26401/1111; 2013-001883-51 (EudraCT Number)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Cognitive Impairment
Keywords: Irdabisant; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — 6-(4-(3-(2-methylpyrrolidin-1-yl)propoxy)phenyl)-2H-pyridazin-3-one; Donepezil; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CEP-26401 5 μg, 25 μg, 125 μg, placebo (Experimental): Participants are dosed four times during this cross-over study. This group takes three active interventions (CEP-26401 in each of the dose options: 5, 25 and 125 μg, and one dose that only contains the placebos.)
  Interventions: Drug: CEP-26401; Drug: Placebo
- CEP-26401 5 μg, 25 μg, placebo, donepezil (Experimental): Participants are dosed four times during this cross-over study. This group takes three active interventions (CEP-26401 at 5 and 25 μg, and donepezil at 10mg and one dose that only contains the placebos.)
  Interventions: Drug: CEP-26401; Drug: donepezil hydrochloride; Drug: Placebo
- CEP-26401 5 μg, 125 μg, placebo, modafinil (Experimental): Participants are dosed four times during this cross-over study. This group takes three active interventions (CEP-26401 at 5 and 125 μg, and modafinil at 200mg) and one dose that only contains the placebos.)
  Interventions: Drug: CEP-26401; Drug: modafinil; Drug: Placebo

INTERVENTIONS:
Drug: CEP-26401 — CEP-26401 as an oral solution at the assigned dose of 5, 25 and/or 125 μg.
  Other Names: Irdabisant
Drug: donepezil hydrochloride — Donepezil hydrochloride, two 5 mg tablets, each over-encapsulated
  Other Names: Aricept
  Arms: CEP-26401 5 μg, 25 μg, placebo, donepezil
Drug: modafinil — modafinil 200 mg tablet, over-encapsulated
  Other Names: Provigil
  Arms: CEP-26401 5 μg, 125 μg, placebo, modafinil
Drug: Placebo — Placebos formulated to match each active drug

SUMMARY:
This is a single center, double-blind, placebo and positive-controlled, randomized, partial 6-way cross-over study to investigate the pharmacodynamics and pharmacokinetics of CEP-26401 (5, 25, and 125 μg) following single-dose administration to healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to give legal informed consent and understand the requirements of the study and communicate with the investigator in the local spoken language.
2. The subject is willing to comply with the study requirements (eg, all dietary, exercise, tobacco, and alcohol restrictions) and provide their written informed consent to participate in the study.
3. The subject is a man or woman, 18 to 50 years of age, inclusive.
4. The subject has a body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive.
5. The subject has skin type I to IV (very light to olive).
6. The subject is in a good health as determined by medical history, ECG, vital signs, physical examination, and clinical laboratory tests.
7. Female subjects of childbearing potential must have a negative serum β-human chorionic gonadotropin (hCG) test (at screening) and check-in and be willing and able to use one of the protocol-specified double-barrier methods of birth control.
8. The subject is able to complete the screening process within 4 weeks prior to study drug administration.

Exclusion Criteria:

1. The subject has a cognitive performance outside of reference values at screening.
2. The subject smokes, is a tobacco user, currently uses nicotine products.
3. The subject has a known hypersensitivity to donepezil, modafinil, irdabisant, or one of the excipients, or has any significant food or drug allergies.
4. The subject is a female who is pregnant or lactating.
5. The subject has an intraocular pressure greater than 22 mm Hg.
6. The subject is suffering from, or has a clinically significant history of one or more of the following: cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s), or a history of any illness that, in the opinion of the investigator, might pose additional risk to the subject by participation in the study or confound the results of the study.
7. The subject has a laboratory abnormality judged by the investigator as clinically significant, or measurements outside of the defined range

   * Other exclusion criteria apply; please contact the investigator for more information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Paired Associate Learning (PAL) Test | Baseline to Hour 22
Rapid Visual Information Processing (RVIP) Test | Baseline to Hour 22
Spatial Working Memory Test | Baseline to Hour 22
Stop Signal Task (SST) | Baseline to Hour 22
Adaptive tracking Test | Baseline to Hour 22
Body sway Test | Baseline to Hour 22
Leeds Sleep Evaluation Questionnaire (LSEQ) | Baseline to Hour 22
Leiden Maze Test (LMT) | Baseline to Hour 22
n-Back Working Memory Test | Baseline to Hour 22
Polysomnography (PSG) Test | Baseline to Hour 22
Saccadic Eye Movements | Baseline to Hour 22
Single-Choice Reaction Time | Baseline to Hour 22
Smooth Pursuit Eye Movements | Baseline to Hour 22
Visual Analog Scales (VAS) | Baseline to Hour 22
  Factors ranging from 'not at all' to 'extremely' are used to quantify subjective drug effects

SECONDARY OUTCOMES:
area under the drug concentration-time curve (AUC0-t) | Baseline to Hour 22
maximal observed plasma drug concentration (Cmax) | Baseline to Hour 22
time to maximum observed plasma drug concentration (tmax) | Baseline to Hour 22
Summary of participants with Adverse Events | From signing of the consent form to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Investigational Site 38051, Leiden, Netherlands